CLINICAL TRIAL: NCT03767660
Title: Efficacy of Rapamycin (Sirolimus) in the Treatment of Blue Rubber Bleb Nevus Syndrome, Hereditary or Sporadic Venous Malformation
Brief Title: Efficacy of Rapamycin (Sirolimus) in the Treatment of BRBNS, Hereditary or Sporadic Venous Malformation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-1606
Record Dates: First submitted 2018-11-24; First posted 2018-12-06 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Blue Rubber Bleb Nevus Syndrome; Venous Malformation
Keywords: Blue Rubber Bleb Nevus Syndrome; Venous Malformation; Rapamycin (sirolimus); Mammalian target of rapamycin (mTOR) inhibitor; Treatment
MeSH Terms: conditions — Blue rubber bleb nevus syndrome; Hereditary Sensory and Autonomic Neuropathies | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapamycin (Experimental): For children: rapamycin, 1 mg per square meter of body surface area a day, orally, for at least 6 months For adults: rapamycin, 2 mg a day, orally, for at least 6 months
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — For children: rapamycin, 1 mg per square meter of body surface area a day, orally, for at least 6 months For adults: rapamycin, 2 mg a day, orally, for at least 6 months
  Other Names: Sirolimus

SUMMARY:
A prospective, nonrandomized, open-label, single-arm clinical trial to study efficacy of rapamycin (sirolimus) in the treatment of Blue Rubber Bleb Nevus Syndrome, hereditary or sporadic venous malformation

DETAILED DESCRIPTION:
Blue rubber bleb nevus syndrome (BRBNS) and venous malformation are mainly caused by somatic mutation of TEK and PIK3CA, which activates the PI3K/AKT signaling pathway. As an important protein kinase downstream of the PI3K/AKT pathway, mTOR can serve as a potential therapeutic target for BRBNS. Experiments of mice have shown that rapamycin inhibited the progression of venous malformation lesions. There are a few human cases reported using rapamycin treatment. The investigator's study is designed to be a prospective, nonrandomized, open-label, single-arm clinical trial to investigate its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with BRBNS, VMCM, sporadic multiple VM, or large single VM;
* Age and gender are not limited;
* Physical status ECOG 0~3;
* Organ function is good, biochemical examination meets the following conditions: AST ≤ 2.5 × upper limit of normal value (ULN), ALT ≤ 2.5 × upper limit of normal value (ULN), serum total bilirubin ≤ 1.5 × upper limit of normal value (ULN), creatinine ≤ 1.5 × upper limit of normal (ULN);
* Patients volunteer to participate in the trial and sign the informed consent form by the participant or his/her legal guardian.

Exclusion Criteria:

* Patients need emergency surgery due to intestinal obstruction, intussusception, or gastrointestinal bleeding;
* History of surgery within 1 month;
* allergic to rapamycin;
* Any disease or condition that may affect the study implementation or result interpretation, including: known hemoglobinopathy, suffering from gastrointestinal infections at the same time, severe heart, liver, kidney and other serious concomitant diseases that may endanger lives
* Pregnant or lactating women;
* Alcohol or drugs (eg, laxatives) abusers;
* Participating in another clinical trial that may affect this study within one month;
* Being believed not suitable to be enrolled by the investigator for other reasons.

Exit Criteria:

* An allergic reaction to rapamycin occurs.
* The patient requests withdrawal: at his own discretion or at the request of his legal representative. Subjects may refuse to participate in further studies at any time without reasons. Subjects will not be affected because of such decision.
* Subjects are required to withdraw from the study in certain special circumstances (eg, there is significant issues of compliance, safety, or surgical intervention for the disease)
* Other situations in which the study must be terminated. For example, the investigators believe that continuing the study may be harmful to the health of subjects.

Rejection Criteria:

* Patients who violate the requirements of the test protocol
* Patients with poor recording (with incomplete, or inaccurate data)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Total venous malformation lesion load | The time from start of therapy to 1 year
  lesion load (cm2) = A + B + C. A = sum of the product of maximum diameter and maximum height of the largest 3 lesions shown by chest, abdomen and pelvis MRI or small bowel CT reconstruction (in cm2) B = sum of the product of maximum diameter and maximum height of the largest 3 lesions shown by digestive endoscope (in cm2) C = sum of the product of maximum diameter and maximum height of the largest 3 lesions shown by ultrasound (in cm2) Remarks: 1. If it is impossible to evaluate 3 or more lesions, results of the actual number of lesions should be taken as valid; 2. Lesions evaluated should be correspondent before and after treatment. If the lesion is difficult to assess after treatment, it should be ruled out from the assessment.

SECONDARY OUTCOMES:
Amount of daily oral iron supplements | The time from start of therapy to 1 year
  The value indicates the amount of gastrointestinal bleeding.
Concentration of hemoglobin in blood | The time from start of therapy to 1 year
  The value indicates the amount of gastrointestinal bleeding.
Frequency of blood transfusion | The time from start of therapy to 1 year
  The value indicates the amount of gastrointestinal bleeding
Concentration of D-dimer in blood | The time from start of therapy to 1 year
  The value indicates the extent of local coagulation caused by Venous Malformation lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Soblet J, Kangas J, Natynki M, Mendola A, Helaers R, Uebelhoer M, Kaakinen M, Cordisco M, Dompmartin A, Enjolras O, Holden S, Irvine AD, Kangesu L, Leaute-Labreze C, Lanoel A, Lokmic Z, Maas S, McAleer MA, Penington A, Rieu P, Syed S, van der Vleuten C, Watson R, Fishman SJ, Mulliken JB, Eklund L, Limaye N, Boon LM, Vikkula M. Blue Rubber Bleb Nevus (BRBN) Syndrome Is Caused by Somatic TEK (TIE2) Mutations. J Invest Dermatol. 2017 Jan;137(1):207-216. doi: 10.1016/j.jid.2016.07.034. Epub 2016 Aug 9. PMID 27519652
- [Background] Ochiai D, Miyakoshi K, Yakubo K, Fukuiya T, Yoshimura Y. Familial blue rubber bleb nevus syndrome in pregnancy with spinal epidural involvement. Case Rep Obstet Gynecol. 2013;2013:141506. doi: 10.1155/2013/141506. Epub 2013 May 9. PMID 23762681
- [Background] Carvalho S, Barbosa V, Santos N, Machado E. Blue rubber-bleb nevus syndrome: report of a familial case with a dural arteriovenous fistula. AJNR Am J Neuroradiol. 2003 Oct;24(9):1916-8. PMID 14561629
- [Background] Kisu T, Yamaoka K, Uchida Y, Mori H, Nakama T, Hisatsugu T, Miyaji H, Motooka M. A case of blue rubber bleb nevus syndrome with familial onset. Gastroenterol Jpn. 1986 Jun;21(3):262-6. doi: 10.1007/BF02774569. PMID 3732758
- [Background] Jin XL, Wang ZH, Xiao XB, Huang LS, Zhao XY. Blue rubber bleb nevus syndrome: a case report and literature review. World J Gastroenterol. 2014 Dec 7;20(45):17254-9. doi: 10.3748/wjg.v20.i45.17254. PMID 25493043
- [Background] Dobru D, Seuchea N, Dorin M, Careianu V. Blue rubber bleb nevus syndrome: case report and literature review. Rom J Gastroenterol. 2004 Sep;13(3):237-40. PMID 15470538
- [Background] Boscolo E, Limaye N, Huang L, Kang KT, Soblet J, Uebelhoer M, Mendola A, Natynki M, Seront E, Dupont S, Hammer J, Legrand C, Brugnara C, Eklund L, Vikkula M, Bischoff J, Boon LM. Rapamycin improves TIE2-mutated venous malformation in murine model and human subjects. J Clin Invest. 2015 Sep;125(9):3491-504. doi: 10.1172/JCI76004. Epub 2015 Aug 10. PMID 26258417
- [Background] Cardoso H, Dias JA, Silva M, Vilas-Boas F, Trindade E, Tavares M, Macedo G. 'Education and Imaging. Gastrointestinal: Successful treatment with sirolimus of a patient with blue rubber bleb nevus syndrome. J Gastroenterol Hepatol. 2016 Mar;31(3):519. doi: 10.1111/jgh.13178. No abstract available. PMID 26456887
- [Background] Yuksekkaya H, Ozbek O, Keser M, Toy H. Blue rubber bleb nevus syndrome: successful treatment with sirolimus. Pediatrics. 2012 Apr;129(4):e1080-4. doi: 10.1542/peds.2010-3611. Epub 2012 Mar 5. PMID 22392180
- [Background] Unlusoy Aksu A, Sari S, Egritas Gurkan O, Dalgic B. Favorable Response to Sirolimus in a Child With Blue Rubber Bleb Nevus Syndrome in the Gastrointestinal Tract. J Pediatr Hematol Oncol. 2017 Mar;39(2):147-149. doi: 10.1097/MPH.0000000000000681. PMID 27820137
- [Background] Salloum R, Fox CE, Alvarez-Allende CR, Hammill AM, Dasgupta R, Dickie BH, Mobberley-Schuman P, Wentzel MS, Chute C, Kaul A, Patel M, Merrow AC, Gupta A, Whitworth JR, Adams DM. Response of Blue Rubber Bleb Nevus Syndrome to Sirolimus Treatment. Pediatr Blood Cancer. 2016 Nov;63(11):1911-4. doi: 10.1002/pbc.26049. Epub 2016 Jun 8. PMID 27273326
- [Background] Moavero R, Coniglio A, Garaci F, Curatolo P. Is mTOR inhibition a systemic treatment for tuberous sclerosis? Ital J Pediatr. 2013 Sep 17;39:57. doi: 10.1186/1824-7288-39-57. PMID 24044547
- [Background] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Background] Paul E, Thiele E. Efficacy of sirolimus in treating tuberous sclerosis and lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):190-2. doi: 10.1056/NEJMe0707153. No abstract available. PMID 18184966
- [Background] Bissler JJ, McCormack FX, Young LR, Elwing JM, Chuck G, Leonard JM, Schmithorst VJ, Laor T, Brody AS, Bean J, Salisbury S, Franz DN. Sirolimus for angiomyolipoma in tuberous sclerosis complex or lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):140-51. doi: 10.1056/NEJMoa063564. PMID 18184959
- [Background] Davies DM, de Vries PJ, Johnson SR, McCartney DL, Cox JA, Serra AL, Watson PC, Howe CJ, Doyle T, Pointon K, Cross JJ, Tattersfield AE, Kingswood JC, Sampson JR. Sirolimus therapy for angiomyolipoma in tuberous sclerosis and sporadic lymphangioleiomyomatosis: a phase 2 trial. Clin Cancer Res. 2011 Jun 15;17(12):4071-81. doi: 10.1158/1078-0432.CCR-11-0445. Epub 2011 Apr 27. PMID 21525172
- [Background] Davies DM, Johnson SR, Tattersfield AE, Kingswood JC, Cox JA, McCartney DL, Doyle T, Elmslie F, Saggar A, de Vries PJ, Sampson JR. Sirolimus therapy in tuberous sclerosis or sporadic lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):200-3. doi: 10.1056/NEJMc072500. No abstract available. PMID 18184971

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT03767660/Prot_SAP_000.pdf